CLINICAL TRIAL: NCT05277480
Title: Apatinib in Combination With Ifosfamide and Etoposide (IE) for Relapsed or Refractory Osteosarcoma Progressed Upon First-line Chemotherapy (AIEO): a Prospective, Multiple-centre, Two-arm, Phase 2 Trial
Brief Title: Apatinib With Ifosfamide Plus Etoposide for Relapsed or Refractory Osteosarcoma (OAIE)
Acronym: OAIE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xie Lu, Musculoskeletal Tumor Center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 11
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Effect of Drug; Drug; Toxicity
Keywords: Osteosarcoma; Apatinib; Ifosfamide; Etoposide
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib+IE group (Experimental): IE: Ifosfamide Plus Etoposide
  Interventions: Drug: Apatinib+IE
- IE group (Active Comparator): IE: Ifosfamide Plus Etoposide
  Interventions: Drug: IE

INTERVENTIONS:
Drug: Apatinib+IE — apatinib po； ifosfamide ivgtt ; etoposide ivgtt .
  Arms: Apatinib+IE group
Drug: IE — ifosfamide ivgtt ; etoposide ivgtt .
  Arms: IE group

SUMMARY:
Apatinib has led to positive responses in the treatment of osteosarcoma refractory to first-line chemotherapy. However, apatinib demonstrates only short-lived activity, and the disease control of musculoskeletal lesions is worse than that of pulmonary lesions. This treatment failure has been partly overcome by the addition of ifosfamide and etoposide (IE). We have ever retrospectively compared the activity of apatinib + IE in relapsed or refractory osteosarcoma in two sarcoma centers in China and concluded that for osteosarcoma with multiple sites of metastasis, apatinib + IE demonstrated clinically meaningful antitumor activity and delayed disease progression in patients with recurrent or refractory osteosarcoma after failure of chemotherapy. However to overcome the influence of other interventions on the outcome, we are currently performing a prospective trial to investigate this combination, from which more accurate data on this treatment strategy are expected.

ELIGIBILITY:
Inclusion Criteria:

1. advanced recurrent and refractory osteosarcoma confirmed by histopathology;
2. initial treatment in the Orthopedic/Oncology Departments of Peking University People's Hospital or Peking University Shougang Hospital;
3. progression less than 6 months after first-line chemotherapy with a combination of high-dose methotrexate, doxorubicin, cisplatin and ifosfamide (first-line chemotherapy);
4. measurable lesions according to the Response Evaluation Criteria for Solid Tumors (RECIST 1.1) ;
5. Eastern Cooperative Oncology Group performance status ≤ 1 ;
6. acceptable haematologic, hepatic, and renal function.

Exclusion Criteria:

1. those who had been previously treated with antiangiogenic TKIs and single IE chemotherapy;
2. those who had severe or uncontrolled medical disorders that could jeopardize the outcomes of the study. These confounding conditions included, cardiac clinical symptoms or disease with left ventricular ejection fraction<50%, and hypertension that could not be well controlled with antihypertensive drugs.;
3. all patients were assessed by the sarcoma board including a thoracic surgeon with at least 10 years surgical experience. Patients with lung metastases only were carefully assessed for eligibility for metastasectomy, of whom those who were suitable for surgery were excluded from this study;
4. weight loss of 20% or more before illness;
5. brain or leptomeningeal metastasis;
6. surgical procedure or radiotherapy within 4 weeks of enrollment;
7. activegastroduodenal ulcer, previous condition associated with risk of bleeding or requiring anticoagulation;
8. proteinuria or hematuria, denutrition with albuminemia <25 g/L;
9. women who were pregnant or breast feeding, other malignancy;
10. positive HBV/HCV/HIV serology, and known allergy to the experimental agents.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-26 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  from the start of target treatment until disease progression or death, whichever came first.

SECONDARY OUTCOMES:
Overall survival | 3 years
  from the date of treatment initiation to death from any cause.

OTHER OUTCOMES:
Objective response rate | 2 years
  defined as the proportion of subjects whose best overall response (BOR) is CR or PR, evaluated by investigator based on RECIST v1.1
Disease control rate | 2 years
  defined as the proportion of subjects whose best overall response (BOR) is complete response (CR), partial response (PR) and stable disease (SD), evaluated by investigator based on RECIST v1.1.
Duration of response | 2 years
  defined as the time from first unconfirmed complete response (CR)/ unconfirmed partial response (PR), evaluated by investigator based on RECIST v1.1, to progressive disease (PD) or any cause of death, whichever occurs first.
Time to response | 2 years
  defined as the time from randomization to first CR/PR, evaluated by investigator based on RECIST v1.1.
Time to progress | 2 years
  defined as the time from randomization to progress disease, evaluated by nvestigator based on RECIST v1.1
Progression-free survival at 4 months | 2 years
  defined as the percentage of patients who were alive and free of disease progression at 4 months evaluated by investigator based on RECIST v1.1
Progression-free survival at 6 months | 2 years
  defined as the percentage of patients who were alive and free of disease progression at 6 months evaluated by investigator based on RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu
  - Shanghai General Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No